CLINICAL TRIAL: NCT04733196
Title: Randomised Controlled Trial Comparing the Clinical Effectiveness of 5 Mouthwashes Based on Essential Oils, Chlorhexidine, Hydrogen Peroxide and Prebiotic, in Gingivitis Treatment
Brief Title: Clinical Effectiveness of 5 Different Mouthwashes in the Treatment of Generalised Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Principal Investigator, Blagovesta Yaneva, Principle investigator, Plovdiv Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PlovdivMU-mouthwash
Record Dates: First submitted 2021-01-22; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Gingivitis
Keywords: Gingivitis; Mouthwashes; Essential oils; chlorhexidine gluconate; hydrogen peroxide; prebiotics; chlorhexidine
MeSH Terms: conditions — Gingivitis | interventions — Oils, Volatile; Prebiotics

STUDY DESIGN:
Intervention Model Description: 180 participants are assigned to 6 groups. Each group of 30 participants with gingivitis rinse with one of the mouthwashes: based on prebiotic, hydrogen peroxide, essential oils, essential oils in combination with 0,12% chlorhexidine, 0,20% chlorhexidine for 3 weeks after mechanical plaque control.
Who Masked: Participant, Care Provider
Masking Description: Participants and providers did not have information about the ingredients in the mouthwashes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Essential oils (Experimental): Mouthwash based on essential oils - menthol, eucalypts oil, thymol, alcohol
  Interventions: Drug: Essential oils
- Essential oils in combination with clorhexidine 0,12% (Experimental): Mouthwash based on essential oils - mentol, eucalypt oil, thymol, alcohol, and 0,12% chlorhexidine
  Interventions: Drug: Essential oils in combination with chlorhexidine 0,12%
- Placebo mouthwash (Placebo Comparator): Water, colorant, sweetener
  Interventions: Drug: Placebo mouthwash
- Clorhexidine 0,20% in combination with aroma oils (Experimental): Mouthwash based on 0,20% chorhexidine without alcohol in combination with aroma oils of rose and lavender
  Interventions: Drug: Chlorhexidine 0,20 % in combination with aroma oils
- Prebiotic (Experimental): Mouthwash based on prebiotic
  Interventions: Drug: Prebiotic
- Hydrogen peroxide (Experimental): Mouthwash based on 0,8% hydrogen peroxide in combination with menthol and eucalypts oil
  Interventions: Drug: Hydrogen peroxide 0,8 %

INTERVENTIONS:
Drug: Essential oils — Participants were asked to rinse with 15 ml mouthwash twice daily for 21 days.
  Arms: Essential oils
Drug: Essential oils in combination with chlorhexidine 0,12% — Participants were asked to rinse with 15 ml mouthwash twice daily for 21 days.
  Arms: Essential oils in combination with clorhexidine 0,12%
Drug: Placebo mouthwash — Participants were asked to rinse with 15 ml mouthwash twice daily for 21 days.
  Arms: Placebo mouthwash
Drug: Chlorhexidine 0,20 % in combination with aroma oils — Participants were asked to rinse with 15 ml mouthwash twice daily for 21 days.
  Arms: Clorhexidine 0,20% in combination with aroma oils
Drug: Prebiotic — Participants were asked to rinse with 15 ml mouthwash twice daily for 21 days.
  Arms: Prebiotic
Drug: Hydrogen peroxide 0,8 % — Participants were asked to rinse with 15 ml mouthwash twice daily for 21 days.
  Arms: Hydrogen peroxide

SUMMARY:
The aim of the present study is to evaluate the efficacy of 5 mouthwashes, based on different ingredients, in the treatment of generalised gingivitis.

DETAILED DESCRIPTION:
The present clinical study aims to investigate the clinical efficacy of 5 mouthwashes based on different active substances. The study include 180 patients divided into 6 groups of 30 patients, each group rinse with one of the following mouthwashes - mouthwash based on essential oils (menthol, thymol and eucalyptus), mouthwash based on essential oils (menthol, thymol and eucalyptus) and 0.12% chlorhexidine, mouthwash based on 0,8 % hydrogen peroxide, mouthwash based on prebiotic, water based on 0.2% chlorhexidine, placebo mouthwash. Inclusion criteria are: generalized gingival inflammation, plaque index of Turesky, 1970 > 1.95, gingival index of Loe & Silness, 1963 > 0.95, no systemic diseases, no systemic medication, lack of severely damaged teeth, no large fillings, no orthodontic treatment. Patients are motivated and instructed to maintain proper and optimal personal oral hygiene. All participants undergo professional mechanical plaque removal. After instrumentation participants are instructed to rinse with 15 ml mouthwash 2 times a day for 21 days. Researchers control the amount of mouthwash used by giving a new bottle of mouthwash with the required amount for 1 patient for 1 week at the beginning of each week and taking back the bottle from the previous week. During the study period, patients are monitored on days 14 and 21, examining plaque index of Turesky, 1970, gingival index of Loe & Silness, 1963, bleeding index of Ainamo & Bay, 1975, side effects like staining, burning itching, oral lesions. At the end of the study (day 21), patients complete a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Plaque Index (Turesky, 1970) > 1,95;
* Gingival Index (Loe & Silness, 1963) > 0,95;
* Bleeding Index (Animo & Bay, 1975) > 30 %;
* no systemic diseases;
* no systemic medication.

Exclusion Criteria:

* severely destroyed teeth;
* crowns;
* non correct obturation class II and V;
* orthodontic treatment;
* third molars.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline bleeding index at 21 day. | 21 days
  Recording the bleeding index of Ainamo&Bay, 1975. The index reports the presence or absence of bleeding on probing in 4 sites around every tooth. It is calculated in % for the whole dentition.

SECONDARY OUTCOMES:
Change from baseline gingival index at 21 day. | 21 days
  The gingival index of Loe, 1967 estimates the inflammation of the gingiva in 4 sites around every tooth, examining the colour, the texture, the consistency and the bleeding of the gingiva.
Change from baseline oral hygiene index at 21 day. | 21 days
  The index of Turesky, 1970 is used. After discolouration of the plaque its distribution is measured in 6 sites of every tooth. The mean value is calculated by summing the individual values for each tooth and dividing the sum by all the places examined.

CONTACTS AND LOCATIONS:
Overall Officials: Blagovesta Yaneva, PhD, Principal Investigator — Plovdiv Medical University
Locations (1):
- Blagovesta Yaneva, Plovdiv, Bulgaria